CLINICAL TRIAL: NCT06309641
Title: Methemoglobinemia Following Intravenous Iron Treatment Administered as Ferric Carboxymaltose or Ferric Derisomaltose in Patients With Anemia
Brief Title: Methemoglobinemia Following Intravenous Iron Treatment
Status: Completed | Type: Observational
Sponsor: Claudia Seiler (Other)
Responsible Party: Sponsor-Investigator, Claudia Seiler, Dr. Claudia Seiler, MD. Consultant anesthesiologist, department of anesthesiology and intensive care medicine Falun hospital, Dalarna County Council, Sweden
Organization: Dalarna County Council, Sweden (Other)
Other Study IDs: MetHb 001
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Methemoglobinemia; Anemia; Iron Deficiencies; Side Effect
Keywords: Intravenous iron; ferric carboxymaltose; ferric derisomaltose
MeSH Terms: conditions — Methemoglobinemia; Anemia; Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ferric derisomaltose: Adult patients with anemia scheduled for administration of ferric derisomaltose as prescribed in routine care.
  Interventions: Diagnostic Test: Blood sample after treatment
- Ferric carboxymaltose: Adult patients with anemia scheduled for administration of ferric carboxymaltose as prescribed in routine care.
  Interventions: Diagnostic Test: Blood sample after treatment
- Case reports: Patients with severe anemia who developed methemoglobinemia after intravenous administration of ferric derisomaltose.
  Interventions: Other: Case reports

INTERVENTIONS:
Diagnostic Test: Blood sample after treatment — Blood samples for measurement of methemoglobin are obtained directly before and 30-120 minutes after drug administration.
  Groups: Ferric carboxymaltose; Ferric derisomaltose
Other: Case reports — Description of clinical course and methemoglobin levels in patients with severe anemia who developed methemoglobinemia after intravenous administration of ferric derisomaltose.
  Groups: Case reports

SUMMARY:
Methemoglobinemia as a side effect of treatment with intravenous iron has not previously been described. This study aims to assess methemoglobin levels in patients with anemia following treatment with intravenous iron, administered as ferric carboxymaltose or ferric derisomaltose.

DETAILED DESCRIPTION:
Methemoglobin is an isoform of hemoglobin without oxygen carrying properties. Higher levels of methemoglobin may impact oxygen transport of the blood and increase the risk of tissue hypoxia. Methemoglobinemia has been reported as side effect of different drugs such as antibiotics or local anesthetics, but not after iron preparations. There is only one case report of increased levels of methemoglobin following intravenous iron therapy.

Patients with anemia due to iron deficiency can be treated with intravenous iron preparations such as ferric carboxymaltose or ferric derisomaltose. Anemia itself reduces oxygen transport of the blood, increasing the risk of tissue hypoxia due to methemoglobinemia in those patients.

This study aims to assess methemoglobinemia following treatment with intravenous iron in patients with anemia. The report will include case reports of patients with severe anemia who developed methemoglobinemia following treatment with ferric derisomaltose. Furthermore, methemoglobin levels are evaluated before and after intravenous iron administration in a cohort of adult patients with anemia who are scheduled to receive ferric carboxymaltose or ferric derisomaltose in routine care.

ELIGIBILITY:
Inclusion Criteria:

for patients in the cohort study:

* anemia
* prescription of administration of intravenous iron (ferric carboxymaltose or ferric derisomaltose)

for patients in the case report:

- patients with severe anemia who developed methemoglobinemia following administration of ferric derisomaltose

Exclusion Criteria:

* declined consent
* known or suspected methemoglobinemia of genetic or other origin
* previous administration of intravenous iron within one week before study sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults (age ≥ 18 years) with anemia that are scheduled for administration of intravenous iron (ferric carboxymaltose or ferric derisomaltose) in the region of Dalarna, Sweden.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Difference in methemoglobin after ferric derisomaltose | 30-120 minutes after start of iron administration
  Change of methemoglobin (percent) in venous blood after compared to before treatment with ferric derisomaltose.
Difference in methemoglobin after ferric carboxymaltose | 30-120 minutes after start of iron administration
  Change of methemoglobin (percent) in venous blood after compared to before treatment with ferric carboxymaltose.

SECONDARY OUTCOMES:
Difference in methemoglobin depending on drug dosage | 30-120 minutes after start of iron administration
  Change of methemoglobin (percent) in venous blood after compared to before treatment with intravenous iron depending on drug dosage
Difference in methemoglobin depending on age | 30-120 minutes after start of iron administration
  Change of methemoglobin (percent) in venous blood after compared to before treatment with intravenous iron depending on age.
Difference in methemoglobin depending on sex | 30-120 minutes after start of iron administration
  Change of methemoglobin (percent) in venous blood after compared to before treatment with intravenous iron depending on sex.
Difference in methemoglobin depending on hemoglobin level before treatment | 30-120 minutes after start of iron administration
  Change of methemoglobin (percent) in venous blood after compared to before treatment with intravenous iron depending on hemoglobin level before treatment.
Difference in methemoglobin depending on blood levels of ferritin, transferrin or iron. | 30-120 minutes after start of iron administration
  Change of methemoglobin (percent) in venous blood after compared to before treatment with intravenous iron depending on blood levels of ferritin, transferrin or iron.
Association between difference in methemoglobin and venous lactate | 30-120 minutes after start of iron administration
  Association between change of methemoglobin (percent) in venous blood and change of lactate in venous blood after compared to before treatment with intravenous iron.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Clinical Research Dalarna, Falun, Sweden